CLINICAL TRIAL: NCT02236598
Title: The Effects of Potassium on Glucose Metabolism in African Americans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00056374
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Borderline Hypokalemia
Keywords: borderline hypokalemia; glucose tolerance; insulin secretion; insulin sensitivity; fasting glucose; African American
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- K+ supplementation (Experimental): K-supplement- Klor-Con® M10 is an immediately dispersing extended-release oral dosage form of potassium chloride containing 750 mg of microencapsulated potassium chloride, United States Pharmacopeia (USP) equivalent to 10 milliequivalent (mEq) of potassium in a tablet. Participants will be instructed to take two 10 mEq tablets twice daily in a blinded encapsulated form, for 3 months
  Interventions: Drug: K+ supplement
- Placebo (Experimental): Placebo - An inert powdered placebo will be identically encapsulated as the Klor-Con intervention tablets to maintain blinding. Participants will be instructed to take two tablets twice daily in a blinded encapsulated form, for 3 months
  Subjects will be instructed to take the pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K+ supplement
  Arms: K+ supplementation
Drug: Placebo
  Arms: Placebo

SUMMARY:
African Americans suffer a disproportionately high risk of diabetes compared to other Americans. Reasons for race disparities in diabetes incidence are not completely understood. Although a difference in prevalence of obesity does explain a significant portion of the racial disparity in diabetes risk, it does not explain all of this disparity. Strategies to control the diabetes epidemic and reduce its racial disparity often overlook preventive measures. Currently, the most powerful known strategy for preventing diabetes is weight loss in the overweight/obese. However, because weight loss is often difficult to achieve and maintain, other opportunities to prevent diabetes should be identified, particularly in African Americans. Among potential novel opportunities is correction of low or low-normal potassium levels (hypokalemia). In secondary analyses, we have found low-normal potassium (K) to be a novel risk factor for diabetes; and we have found that this association between low-K and diabetes risk may be stronger in African Americans compared to whites. Therefore, a previously unrecognized alternative or adjunct strategy for preventing diabetes, particularly in African Americans, may involve correction of low or low-normal K levels (hypokalemia). Large-scale, adequately-powered, randomized controlled trials are needed to establish the effectiveness of this approach. However, prior to those trials, the pathophysiology of the association between low K and poor glucose metabolism must be understood. This pilot clinical trial will begin to determine the effect of K supplementation on measures of glucose metabolism in African Americans.

In this pilot clinical trial, 30 African Americans with prediabetes and a low-normal serum K [<4.0 milliequivalent/Liter (Eq/L)] will be randomized to K-supplements, 20mEq (2-10mEq tablets) twice daily or a matching placebo capsules twice daily. Prior to randomization, baseline measures will be taken including measures of glucose metabolism with a 3-hour oral glucose tolerance test (OGTT), baseline chemistries and a baseline 24-hour urinary potassium measurement. Patients will take the intervention daily and will undergo repeat testing of all of these measures at the end of a 3 month period. The primary endpoint will be change in glucose tolerance, as measured by change in glucose area-under-the-curve (AUC) of a 3-hour oral glucose tolerance test (OGTT). Secondary endpoints will include changes in fasting, 1-hour, and 2-hour post-challenge glucose levels, as well as measurements of insulin secretion and insulin sensitivity as measures by the oral glucose minimal model method.(1) The baseline data from this trial will allow us to quantify abnormalities in glucose metabolism in African Americans with prediabetes/early diabetes and low-normal serum K. The post-intervention data will provide estimates of the impact of K-supplements compared to no supplements on these abnormalities. Data derived from the pilot study will be used in the design of a larger scale, adequately powered clinical trial. This trial will also help to assess the feasibility of recruiting this target population.

With this pilot trial, we will begin to determine whether or not K-supplements, an inexpensive, well-tolerated, and simple intervention, could help to reduce diabetes risk among African Americans.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in the study the following enrollment criteria must be met:

1. Participants must be 30 years of age or older.
2. They must have a diagnosis of prediabetes defined as a hemoglobin A1c between 5.7-6.5% measured at the initial screening visit.
3. They must have a serum K+ of 3.3-4.0 mEq/L on 2 occasions, within a 18 month period, including at initial screening visit. If subject is just outside range for inclusion, PI may offer the subject the option to repeat their screening serum K+ measurement.
4. The participant must be willing and capable of providing written informed consent.
5. The participant must be available for follow-up and must at minimum have telephone access.
6. Participants must be able to read/understand English.

Exclusion Criteria:

* Participants must not have any of the following:

  1. Participants must not have evidence of chronic kidney disease with an estimated Glomerular Filtration Rate (eGFR) < 60ml/min. All patients will be screened for eGFR at the enrollment visit.
  2. Participants must not have evidence of diabetes mellitus requiring treatment with medications prior to screening visit. The cannot have a random or post-challenge glucose ≥ 200mg/dl (from prior labs), A1c level ≥ 6.5% (from prior labs), prior physician diagnosis, or use of anti-diabetic medications. If participants have glucose levels in the diabetic range at screening visit, they will be eligible to continue in study as long as glucose levels are not > 200 mg/dl.
  3. Participants must not have a history of endoscopy-verified peptic ulcer disease with past history of either gastric or duodenal ulcer.
  4. Participants must not have evidence of cardiac arrhythmias, unstable angina or cardiac event within 6 months, congestive heart failure, or other conditions that might impact follow-up, based on the discretion of the principal investigator.
  5. Participants must not be pregnant or intend to get pregnant during the study period. The study intervention is safe for pregnant women, so serum pregnancy screening is not indicated; however, pregnant women are excluded because pregnancy affects glucose homeostasis, which will bias primary outcome measurement and damage scientific validity of the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranee C Montgomery, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Chatterjee R, Davenport CA, Kwee L, D'Alessio D, Svetkey LP, Lin PH, Slentz CA, Ilkayeva O, Johnson J, Edelman D, Shah SH. Preliminary evidence of effects of potassium chloride on a metabolomic path to diabetes and cardiovascular disease. Metabolomics. 2020 Jun 18;16(7):75. doi: 10.1007/s11306-020-01696-w. PMID 32556595
- [Derived] Chatterjee R, Slentz C, Davenport CA, Johnson J, Lin PH, Muehlbauer M, D'Alessio D, Svetkey LP, Edelman D. Effects of potassium supplements on glucose metabolism in African Americans with prediabetes: a pilot trial. Am J Clin Nutr. 2017 Dec;106(6):1431-1438. doi: 10.3945/ajcn.117.161570. Epub 2017 Nov 1. PMID 29092881

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 61 participants (17%) expressed interested in the study and signed informed consent. Of these, 29 participants were deemed eligible based on the results of the screening labs
Groups:
- K+ Supplementation: K-supplement- Klor-Con® M10 is an immediately dispersing extended-release oral dosage form of potassium chloride containing 750 mg of microencapsulated potassium chloride, USP equivalent to 10 mEq of potassium in a tablet. Participants will be instructed to take two 10 mEq tablets twice daily in a blinded encapsulated form, for 3 months
  K+ supplement
- Placebo: Placebo - An inert powdered placebo will be identically encapsulated as the Klor-Con intervention tablets to maintain blinding. Participants will be instructed to take two tablets twice daily in a blinded encapsulated form, for 3 months
  Subjects will be instructed to take the pills
  Placebo
Period: Overall Study
Arm/Group | K+ Supplementation | Placebo
Started | 15 | 14
Completed | 15 | 12
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 14 participants started in the placebo arm, but only 12 completed and included in the Baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | K+ Supplementation | Placebo | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (11.0) | 52.7 (8.9) | 55.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 27
BMI [Mean (Standard Deviation); unit: kg/m2] | 34.3 (5.4) | 35.1 (5.2) | 34.8 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glucose Tolerance as Measured by Area-under-the-curve
Description: Change in glucose tolerance, as measured by change in glucose area-under-the-curve (Area Under the Curve (AUC) - measured via the trapezoidal method) of 2 hours from the 3-hour Oral Glucose Tolerance Test (OGTT).
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: AUC - mg*min/dL
Arm/Group | K+ Supplementation | Placebo
Number analyzed (Participants) | 15 | 12
AUC - mg*min/dL | 328 (1779) | 1000 (2378)
Statistical Analysis 1: Comparison: K+ Supplementation vs Placebo; Test type: Superiority; p = 0.5582, ANCOVA

2. Secondary Outcome: Changes in Fasting, 1-hour, and 2-hour Post-challenge Glucose Levels in mg/dL
Description: Changes in fasting, 1-hour, and 2-hour post-challenge glucose levels in mg/dL
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | K+ Supplementation | Placebo
Number analyzed (Participants) | 15 | 12
mg/dL
  Change in Fasting Glucose | -1.0667 (8.3961) | 6.0833 (7.6093)
  Change in 1-Hour Glucose | 0.80 (31.36) | 14.17 (37.07)
  Change in 2-Hour Glucose | 3.60 (25.82) | 0.75 (24.53)
Statistical Analysis 1: Comparison: K+ Supplementation vs Placebo; Test type: Superiority — Change in Fasting Glucose; p = 0.0963, ANCOVA
Statistical Analysis 2: Comparison: K+ Supplementation vs Placebo; Test type: Superiority — Change in 1-hour Glucose; p = 0.6671, ANCOVA
Statistical Analysis 3: Comparison: K+ Supplementation vs Placebo; Test type: Superiority — Change in 2-hour Glucose; p = 0.7913, ANCOVA

3. Secondary Outcome: Changes in Insulin Secretion as Measured by 2-hour Insulin Area-under-the-curve (AUC)
Description: Changes in Insulin Secretion as measured by 2-hour insulin area-under-the-curve (AUC - measured via the trapezoidal method) of 2 hours from the 3-hour OGTT.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: AUC - pg*min/mL
Arm/Group | K+ Supplementation | Placebo
Number analyzed (Participants) | 15 | 12
AUC - pg*min/mL | 71,444 (213,221) | 149,327 (378,900)
Statistical Analysis 1: Comparison: K+ Supplementation vs Placebo; Test type: Superiority; p = 0.5294, ANCOVA

4. Secondary Outcome: Changes in Insulin Sensitivity
Description: Matsuda Insulin Sensitivity Index was calculated as: 10,000 / square root of [fasting glucose x fasting insulin x mean glucose x mean insulin during Oral Glucose Tolerance Test]).
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: AUC - unitless,
Arm/Group | K+ Supplementation | Placebo
Number analyzed (Participants) | 15 | 12
AUC - unitless, | -0.03 (1.49) | -0.87 (1.13)
Statistical Analysis 1: Comparison: K+ Supplementation vs Placebo; Test type: Superiority; p = 0.1604, ANCOVA

ADVERSE EVENTS:
Time Frame: The reporting period for SAEs is from the day of randomization and receipt of study medication through 12-week end-of-study visit.
Arm/Group | K+ Supplementation | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | K+ Supplementation (N=15) | Placebo (N=14)
Vasovagal Syncope (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No